CLINICAL TRIAL: NCT06529874
Title: Pressure Pain Tolerance in Relation to Balance and Strength in Children With Sickle Cell Anemia
Brief Title: Pressure Pain Tolerance in Relation to Balance and Strength in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adly A Adam (Other)
Responsible Party: Sponsor-Investigator, Adly A Adam, Lecturer Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/005092
Record Dates: First submitted 2024-07-25; First posted 2024-07-31 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: An observational correlational study design.
Masking Description: Forty normal healthy children from primary governmental schools at Alexandria governate, and Forty children with sickle cell anemia from Alexandria University Students Hospitals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Healthy children (Experimental): All forty normal healthy children will undergo measurement of pressure pain tolerance via digital pressure algometry, balance assessment using HUMAC balance system, and evaluation lower limb strength using Lafayette Hand Held Dynamometer.
  Interventions: Other: Pressure pain tolerance measurement using Digital Pressure Algometer; Other: Balance assessment using HUMAC balance system; Other: Lower limb muscular strength using Lafayette hand held dynamometer
- Sickle cell anemia children (Experimental): All forty Sickle cell anemia children will undergo measurement of pressure pain tolerance via digital pressure algometry, balance assessment using HUMAC balance system, and evaluation lower limb strength using Lafayette Hand Held Dynamometer.
  Interventions: Other: Pressure pain tolerance measurement using Digital Pressure Algometer; Other: Balance assessment using HUMAC balance system; Other: Lower limb muscular strength using Lafayette hand held dynamometer

INTERVENTIONS:
Other: Pressure pain tolerance measurement using Digital Pressure Algometer — Pressure pain tolerance will be measured using pressure algometer for all participants in both groups. Pressure pain tolerance will be measured in a relaxed sitting position to evaluate on quadriceps muscle. Initially, a teddy bear will be used for demonstration.
Other: Balance assessment using HUMAC balance system — HUMAC balance system will be calibrated, then will conduct
  1. center of pressure: will instructed child to stand on platform, and maintain own body stability, and focus on the red dot in the center of screen that will move in response to body sway. after a rest, second trial will be done.
  2. Eye open/ closed firm surface tests: First for Eye open firm surface test; the child will be asked to look at a target on the wall that was set at his/ her eye level, and to stare at this target for 30 seconds while standing on firm surface. After 5 seconds rest. Eye closed firm surface test; child will be asked to close his/ her eyes for 30 seconds, and conducting the same procedures for balance testing.
  The researcher will documented the values resented on the screen .
Other: Lower limb muscular strength using Lafayette hand held dynamometer — Lower limb muscular ' Isometric quadriceps strength' will be measured for all participants in both groups. each participating child will be instructed to sit to assess the strength of knee extension, which minimize positional changes, and enhance feasibility of this clinical test. then The researcher will apply resistance to child's quadriceps to gain maximal voluntary isometric contraction with pressing the activated Lafayette hand held dynamometer padded stirrup against quadriceps belly, then recorded and documented measured value.
  Other Names: Isometric quadriceps strength'

SUMMARY:
Sickle cell disease (SCD) is the most frequent life-threatening genetic hemoglobinopathy in the world and occurs due to the synthesis of abnormal hemoglobin S (HbS).Cells with sickle cell hemoglobin are stiff and sticky. When they lose their oxygen, they form into the shape of a sickle or crescent. This can cause pain and tissue damage. Significant decrease in exercise capacity was seen in sickle cell anemic children. In the absence of a guidelines that can guide the prescription of exercise in SCD children. This study is a step for determine the forms of prescription of pain on the balance and muscle strength to build up in future studies a safety of physical exercises for children with sickle cell anemia and improve their functional abilities.

DETAILED DESCRIPTION:
Sickle cell anemia is a serious life-limiting and potentially life-threatening condition that causes disruption in the lifestyle of the affected child. Pain is a common and severe symptom of sickle cell disease (SCD) and is the major reason that patients seek health care services. Some researchers supported the fact that an important impairment in balance control and muscle strength in children with sickle cell disease due to pressure pain tolerance problems and other factors. Significant decrease in exercise capacity was seen in sickle cell anemic children. The altered muscle function and balance observed in SCD children may collectively be the result of pressure pain tolerance impairment. As your physical fitness improves, your body becomes more efficient at getting oxygen into the bloodstream and transporting it to the working muscles. Along this observational correlational study design; Eighty children from both sexes will be participated in this study. Forty normal healthy children will be selected from primary governmental schools at Alexandria governorate and forty children with sickle cell anemia will be selected from Alexandria University Students Hospitals For evaluation of muscle strength hand held dynamometer (Lafayette) is one of the best methods to detect the muscle strength. It is an ergonomic hand-held device for objectively quantifying muscle strength

ELIGIBILITY:
Inclusion Criteria:

* Age range range was 9-14 years old.
* Could follow given instructions.
* Children with Sickle cell anemia were medically stable, and take their medications regularly.
* Children with Sickle cell anemia had experience of chronic pain that lasts more than 6 months.
* All children with Sickle cell anemia have average weight, height, and body mass index based on their age percentiles.
* All normal healthy children did not participating in regular sport activities, particularly including lower limb strengthening.

Exclusion Criteria:

* Defined cardiovascular or respiratory disorders.
* Renal failure.
* Myocardial infarction, mainly within last month.
* Unstable angina.
* Recent thoracoabdominal surgery.
* Thoracic or abdominal aneurysm or current pneumothorax.
* Painful vaso-occlusive crises.
* Muscular contractures, Joints' stiffness, or deformities.
* Neuromuscular problems i.e., myositis or peripheral neuropathy.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Pressure pain tolerance | Baseline of the study.
  Pressure pain tolerance measured via digital pressure algometer. It determines the pressure amount could be tolerated over quadriceps. This will represented chronic pain among Sickle cell anemia children in order to aid in diagnosis of hyperalgesia thus provide insight into their management strategies. Digital pressure algometer determines enables the rater to quantify the mechanical sensitivity to pain and the recovery of underlying problems or soreness levels in a semi-objective manner.
Balance assessment | Baseline of the study.
  Balance assessed via HUMAC balance system to define musculoskeletal involvement in sickle cell anemia children. HUMAC balance system is an electronic balance board connected with laptop running HUMAC balance system software.
Lower limb muscle strength | Baseline of the study.
  Lower limb muscle (Quadriceps) strength evaluated via Lafayette hand held dynamometer to evaluate voluntary isometric contraction. Hand held dynamometer has a good to excellent reliability and validity mainly for proximal musculatures.

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa A Ahmed, PHD, Study Chair — Head of Haematology Dept, Faculty of Medicine, Alexandria University; Elham M Salem, PHD, Study Director — Professor of Physical Therapy, Faculty of Physical Therapy, Cairo University
Locations (1):
- El-Tahrir st.- in front of Ben El-Sarayat, Ad Doqi Al Giza, Giza Governate, Giza, Egypt